CLINICAL TRIAL: NCT03541564
Title: A Randomized, Double-Blind, Positive-Controlled, Placebo-Controlled, 4-Period Crossover Study to Investigate the Electrocardiographic Effects of BMS-986165 in Healthy Subjects
Brief Title: An Investigational Study of Experimental Medication BMS-986165 in Healthy Participants to Study Electrocardiogram Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-048
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Systemic Lupus Erythematosus; Healthy Participants
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — deucravacitinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986165 Dose 1 oral administration (Experimental): BMS-986165 therapeutic single dose
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 2 oral administration (Experimental): BMS-986165 supratherapeutic single dose
  Interventions: Drug: BMS-986165
- Moxifloxacin Dose 3 oral administration (Active Comparator): Moxifloxacin positive control single dose
  Interventions: Drug: Moxifloxacin
- Placebo Dose 4 oral administration (Placebo Comparator): Placebo single dose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Arms: BMS-986165 Dose 1 oral administration; BMS-986165 Dose 2 oral administration
Drug: Moxifloxacin — Specified dose on specified days
  Arms: Moxifloxacin Dose 3 oral administration
Other: Placebo — Specified dose on specified days
  Arms: Placebo Dose 4 oral administration

SUMMARY:
This is a study to investigate the experimental medication BMS-986165 in healthy participants in order to study the effects it has on electrocardiogram results.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations in the opinion of the investigator
* Body mass index of 18.0 to 32.0 kg/m2, inclusive, and body weight ≥ 50 kg, at screening
* Normal renal function at screening as evidenced by an estimated glomerular filtration rate (GFR) > 80 mL/min/1.732 m2

Exclusion Criteria:

* Any medical condition that presents a potential risk and/or may compromise the objectives of the study, including a history or presence of active liver disease
* A personal history of clinically relevant cardiac disease as determined by the investigator, symptomatic or asymptomatic arrhythmias, presyncope or syncopal episodes, or additional risk factors for torsades de pointes (eg, heart failure)
* History of hypokalemia, personal history or family history of prolonged QT interval, or family history of sudden cardiac death at a young age

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change from baseline in (Fridericia) QT Interval (QTcF) for BMS-986165 as determined by 12-lead electrocardiogram (ECG) | From baseline to 5 days

SECONDARY OUTCOMES:
Placebo-corrected change from baseline in corrected (Fridericia) QT Interval (QTcF) for moxifloxacin as determined by 12-lead ECG | From baseline to 5 days
Heart rate (HR) as determined by 12-lead ECG | 5 days
QRS as determined by 12-lead ECG | 5 days
PR as determined by 12-lead ECG | 5 days
Change from baseline in corrected (Fridericia) QT Interval (QTcF) as determined by 12-lead ECG | From baseline to 5 days
Incidence of participant abnormalities in vital signs, clinical laboratory tests, safety 12-lead ECGs, and physical examinations | Up to 28 days
Incidence of adverse events (AE) | Up to 28 days
Incidence of serious adverse events (SAE) | Up to 28 days
Maximum observed concentration (Cmax) as determined by plasma concentration | 5 days
Time of maximum observed concentration (Tmax) as determined by plasma concentration | 5 days
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] as determined by plasma concentration | 5 days
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] as determined by plasma concentration | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm